CLINICAL TRIAL: NCT06705439
Title: A Study of Detection of Paroxysmal Events Utilizing Computer Vision and Machine Learning (USF)
Status: Recruiting | Type: Observational
Sponsor: Neuro Event Labs Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: STUDY005226
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Epilepsy
Keywords: Nelli
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Nelli — Nelli detects and registers activity that is indicative of seizure events. Nelli captures, stores, and processes video and audio recordings from each patient. Biomarker data is collected during periods of rest for the length of an examination period, which may span several days or months (when used inside and outside of a hospital setting, respectively), as prescribed by a treating physician.

SUMMARY:
Increased computational power has made it possible to implement complex image recognition tasks and machine learning to be implemented in every day usage. The computer vision and machine learning based solution used in this project (Nelli) is an automatic seizure detection and reporting method that has a CE mark for this specific use.

The present study will provide data to expand the utility and detection capability of NELLI and enhance the accuracy and clinical utility of automated computer vision and machine learning based seizure detection.

DETAILED DESCRIPTION:
This is a prospective, blind comparison to the clinical gold standard for seizure characterization. This study is intended to compare the Nelli Software's ability to identify seizure events to vEEG review in adults with suspected nighttime seizures. Simultaneously, Nelli will continuously record audio and video while video-electroencephalography (vEEG) is recorded per typical standard of care. Events with positive motor manifestations will be independently identified, following standard clinical practice, by three epileptologists using clinical vEEG data. Nelli Software will review the audio and video data and independently identify events with positive motor manifestations. The outcomes of event identification will be compared between Epileptologists and the Nelli Software. For each category of event captured the positive percent agreement will be calculated using the exact binomial method. The primary endpoint of this study is to demonstrate that Nelli is able to identify seizures that have a positive motor component with a sensitivity of > 70%.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing video-EEG monitoring for clinical purposes who are suspected of having seizures.

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected motor seizures that are undergoing video-EEG monitoring for routine clinical care.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of a seizure detection system | During routine seizure monitoring in the hospital - up to one week
  The primary outcome measure will be the sensitivity of the Nelli system to detect seizrues with a positive motor component in comparison to independent Neurologist review of vEEG collected in an epilepsy monitoring unit. This is a blinded comparison to the clinical gold standard (vEEG)

CONTACTS AND LOCATIONS:
Overall Officials: Selim Benbadis, MD, Principal Investigator — University of South Florida
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No